CLINICAL TRIAL: NCT06537661
Title: VIRTUAL REALITY and TEMPOROMANDIBULAR DISORDER FOLLOWING MAXILLOFACIAL SURGERY
Brief Title: Effect of Virtual Reality on TMD Following Maxillofacial Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nehal mohamed soliman Elbkery, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005153
Record Dates: First submitted 2024-07-02; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Temporomandibular Disorder
Keywords: VR; TMD; Maxillofacial surgery
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): VR and traditional Ex
  Interventions: Other: Virtual reality
- Control group (Experimental): traditional physical therapy ex
  Interventions: Other: Traditional exercises

INTERVENTIONS:
Other: Virtual reality — Virtual reality (VR): is the artificial construction of a 3D environment viaThe VR glasses which were the source of visual and auditory feedback, were connected by Bluetooth to a mobile phone and all the videos of selected tasks.
  Arms: Study group
Other: Traditional exercises — Active mobility exercises (jaw opening 6 times of 30 s; lateralization 10 times of 5 s; protrusion 10 times Of 5 s). Self-massage masticatory Muscles, After each session.
  * Isometric contraction exercises Were included (3 times of 10 s)
  Arms: Control group

SUMMARY:
Sixty eight patients who have TMJ pain and ROM restriction after maxillofacial surgery participated in this study , they are selected from government hospitals (general and insurance ).

Will be randomly divided into two equal groups ( group A, group B ). Their ages range from 20 - 35 years.

The Purpose of the study is to evaluate the therapeutic efficacy of VR in decreasing pain and improve ROM for Patients after maxillofacial surgery.

DETAILED DESCRIPTION:
Sixty eight patients who have TMJ pain and ROM restriction after maxillofacial surgery participated in this study , they are selected from government hospitals (general and insurance ).

Will be randomly divided into two equal groups ( group A, group B ). Their ages range from 20 - 35 years.

The VR glasses which were the source of visual and auditory feedback, were connected by Bluetooth to a mobile phone and all the videos of selected tasks (tasks of Active mobility exercises and isometric contraction exercises, massage exercises) were turned on. Active mobility exercises (jaw opening 6 times of 30 s; lateralization 10 times of 5 s; protrusion 10 times Of 5 s).

* Self-massage masticatory Muscles, After each session.
* Isometric contraction exercises The Purpose of the study is to evaluate the therapeutic efficacy of VR in decreasing pain and improve ROM for Patients after maxillofacial surgery.

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:

  * Patients after Arthrocentesis .
  * Patients after Temporomandibular joint condylar discopexy.
  * Age ranges between 30 - 45 years.
  * All patients will have informed consent .Exclusion Criteria:
* • Surgery That conducted on the temporomandibular joint (meniscectomy, arthroscopy, etc.).

  * oral surgery (e.g., surgery for impaction of the third molar), as well as patients with concomitant systemic or neurological conditions.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Measure pain | 6weeks
  Measure by visual analog scale (VAS) 0: low in pain 10:high in pain

SECONDARY OUTCOMES:
Maximum mouth opnening (MMO ) | 6weeks
  Measure by milemeter

CONTACTS AND LOCATIONS:
Locations (1):
- Nehal mohamed, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No